CLINICAL TRIAL: NCT02695693
Title: RCT of TeachTown in Autism Support Classrooms: Innovation and Exnovation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The School District of Philadelphia (Other)
Responsible Party: Principal Investigator, David Mandell, Director, Center for Mental Health Policy and Services Research, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH106175 (NIH); R01MH106175 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TeachTown (Experimental): Students in kindergarten-through-second-grade autism support classrooms in this arm receive access to TeachTown, an online academic and pre-academic intervention designed for students with autism. Their teachers also receive coaching in the use of TeachTown, as well as coaching in other evidence-based practices for students with autism, including discrete trial training, pivotal response training, and teaching in functional routines
  Interventions: Behavioral: TeachTown; Behavioral: Discrete Trial Training; Behavioral: Pivotal Response Training; Behavioral: Teaching in Functional Routines
- Control (Active Comparator): Teachers in kindergarten-through-second-grade autism support classrooms in this arm receive coaching in evidence-based practices for students with autism, including discrete trial training, pivotal response training, and teaching in functional routines
  Interventions: Behavioral: Discrete Trial Training; Behavioral: Pivotal Response Training; Behavioral: Teaching in Functional Routines

INTERVENTIONS:
Behavioral: TeachTown — TeachTown is an online program for students with autism that uses an applied behavior analysis framework to provide intervention in academic and pre-academic areas
  Arms: TeachTown
Behavioral: Discrete Trial Training — Discrete trial training is a one-on-one didactic behavioral intervention in which the teacher or therapist uses specific behavioral methods based on principles of operant conditioning, to help students gain skills
Behavioral: Pivotal Response Training — Pivotal response training is a one-on-one child-lead behavioral intervention in which the teacher or therapist uses specific behavioral methods, leveraging the students interests, to help students gain skills
Behavioral: Teaching in Functional Routines — Functional routines are sets of chained behaviors that students are taught that help them complete and manage specific activities in the classroom

SUMMARY:
Computer assisted interventions are becoming very popular as an intervention strategy for students with autism. There is little data on how effective they are or how their implementation affects teachers' use of other evidence-based practices. The proposed study would be the first to examine these questions in a community setting.

DETAILED DESCRIPTION:
This study comprises a randomized controlled trial to examine 1) the effectiveness of TeachTown: Basics, one of the only evidence-based computer-assisted intervention (CAI) packages for students with autism; 2) the extent to which teachers implement TeachTown the way it was designed; 3) the effects of its use on other evidence-based practices; and 4) organizational and teacher variables that mediate changes in the use of evidence-based practices when TeachTown is introduced. While there has been a rush to take advantage of CAI, there is little research on whether it will result in better outcomes for student with autism, and be feasible or sustainable in community settings. While CAI has the potential to increase instructional time for students with autism, it may result instead in teachers reducing their use of other evidence-based practices, including the amount of interpersonal (as opposed to computer) instruction students receive. While the related constructs of exnovation, de-implementation and de-adoption have been used to describe this phenomenon for more than 30 years, they rarely have been systematically studied. The proposed study takes advantage of an ongoing rollout of TeachTown in the School District of Philadelphia. TeachTown includes a computerized instruction component, combined with offline, interpersonal instruction between the student and teacher. It is not known whether public schools have the resources to implement programs like this, regardless of their efficacy, or whether or how teachers will incorporate them into the instructional day. An especially important question is whether existing evidence-based practices are exnovated as TeachTown is implemented. To address these questions, we rely on our longstanding collaboration with the School District of Philadelphia, the 8th largest school district in the US. At the beginning of the school year, we will inventory relevant technology and observe how it is used in the District's 83 kindergarten-through-second-grade autism support classrooms. We also will survey teachers and school administrators about expectations, support and rewards for using these technologies and attitudes, norms and self-efficacy regarding the use of these technologies. We then will use a waitlist-control randomized design to examine TeachTown's effects on student outcomes and use of other practices. We will unpack the impact of the implementation of TeachTown on existing evidence-based practices using direct observation and through qualitative interviews. The waitlist design allows the district to roll out the intervention to all classrooms, which is their intent. It also allows s to increase our sample to study moderators of sustainment of existing EBPs when a new technology is introduced. The proposed study would be one of the first to examine longitudinally the uptake of new technology for children with ASD in school settings, and the first to address use of CAI. Successful completion of this study will identify malleable targets for intervention to increase the use of CAI, should that appear warranted, while sustaining existing EBPs for children with autism in community settings.

ELIGIBILITY:
Inclusion Criteria:

* educational classification of autism, receiving services in a kindergarten-through-second-grade autism support classroom in the School District of Philadelphia, with a teacher who has agreed to participate in the study, and parents speak English or Spanish

Exclusion Criteria:

* none

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Differential Abilities Scale, 2nd Edition | 8 months
  A nationally normed battery of cognitive and achievement tests.
Bracken School Readiness Assessment, 3rd Edition | 8 months
  n individual cognitive test designed for children, pre-K through second grade

REFERENCES:
- [Derived] Pellecchia M, Marcus SC, Spaulding C, Seidman M, Xie M, Rump K, Reisinger EM, Mandell DS. Randomized Trial of a Computer-Assisted Intervention for Children With Autism in Schools. J Am Acad Child Adolesc Psychiatry. 2020 Mar;59(3):373-380. doi: 10.1016/j.jaac.2019.03.029. Epub 2019 Apr 3. PMID 30953731
- [Derived] Pellecchia M, Beidas RS, Marcus SC, Fishman J, Kimberly JR, Cannuscio CC, Reisinger EM, Rump K, Mandell DS. Study protocol: implementation of a computer-assisted intervention for autism in schools: a hybrid type II cluster randomized effectiveness-implementation trial. Implement Sci. 2016 Nov 25;11(1):154. doi: 10.1186/s13012-016-0513-4. PMID 27884169